CLINICAL TRIAL: NCT05621213
Title: Satisfaction of Patients With Amyotrophic Lateral Sclerosis Under Non-invasive Ventilation Regarding Home Assisted Teleconsultation
Brief Title: Satisfaction of Patients With Amyotrophic Lateral Sclerosis Regarding Home Assisted Teleconsultation
Acronym: VNI_SLA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to insufficient recruitment despite mitigation measures, as enrolment rates could not meet protocol objectives. Academic thesis scheduling constraints also contributed. No safety concerns were identified.
Sponsor: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-A01667-36
Record Dates: First submitted 2022-10-27; First posted 2022-11-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: ALS; Charcot Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Nurses

STUDY DESIGN:
Intervention Model Description: Patient assigned to the interventional group or to the control group if they do not wish to be followed up by teleconsultation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients who will be followed up by teleconsultation assisted by a physiotherapist or a nurse at home.
  Interventions: Other: Teleconsultation assisted by a physiotherapist or nurse
- Control group (No Intervention): Patients not wishing to be followed up by teleconsultation but agreeing to participate in the study and the collection of questionnaires. They will follow up as usual in person (no teleconsultation).

INTERVENTIONS:
Other: Teleconsultation assisted by a physiotherapist or nurse — A home health care provider (with expertise in NIV) will be asked to attend the 2 home teleconsultation sessions.
  This assistance will make it possible to help, if necessary, the patient to settle in and connect, collect the elements necessary for the doctor's consultation and adjust, if necessary, the NIV settings. He will also be responsible for administering the questionnaires to the patient as well as to his family caregiver.
  Arms: Intervention

SUMMARY:
Satisfaction of patients with amyotrophic lateral sclerosis under non-invasive ventilation regarding home assisted teleconsultation

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a progressive and rapidly progressing neurodegenerative disease. Depending on the degree of muscle damage, patients may suffer from reduced mobility, difficulty swallowing, speech difficulties and finally respiratory weakness. Death occurs within an average of 2-3 years and is usually due to respiratory failure. Currently there is no cure for ALS, so palliative care and symptomatic treatments are essential for the management of these patients.

The gold standard treatment for respiratory impairment is non-invasive ventilation (NIV). The aim of this mask ventilation is to improve gas exchange by compensating for the weakness of the respiratory muscles.

The progressive nature of ALS requires regular assessment of the patient's clinical condition and evaluation of NIV parameters. Regular medical appointments are therefore essential to ensure optimal ventilation and close surveillance of the patient. A day hospitalization or a consultation is organized every 3 or 4 months. These visits can cause significant fatigue, not only because of the difficulty patients have to move around but also because of the time spent waiting in hospital.

ALS is characterised by its severity and it requires our society to think about and implement new ways of managing the disease. Thus, e-health innovations could be an interesting potential in the remote follow-up of these patients, to reduce the burden of hospital consultations.

The hypothesis is that the patient will be more satisfied with a home assisted teleconsultation follow-up, while keeping the same quality of non-invasive nocturnal ventilatory assistance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of ALS coming for a follow-up consultation with their pneumologist
* Daily NIV compliance of more than 4 hours in the month prior to inclusion
* Living at home
* Patient with a natural caregiver
* Patient equipped with computer equipment adapted for teleconsultation (tablet, computer, telephone... with an internet connection)
* Patient able to read and understand the procedure, and able to express consent for the study protocol
* Patient, or his or her caregiver, able to sign the consent to participate by himself or herself

Exclusion Criteria:

* Patient not available or wishing to change region within 3 months of inclusion
* Patient currently participating or having participated in the month prior to inclusion in another clinical interventional research study that may have an impact on the study, this impact is left to the discretion of the investigator
* Persons referred to in articles L1121-5 to L1121-8 of the French Public Health Code (corresponding to all protected persons)
* Pregnant women (for women of childbearing age and in the absence of reliable contraception, the β-HCG (human chorionic gonadotropin) assay will be performed), parturient women, breastfeeding women,
* persons deprived of their liberty by judicial or administrative decision,
* persons under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Satisfaction of ALS patients followed by teleconsultation at home | Between the initial visit and the 3-month visit
  Evolution of the overall satisfaction score obtained from the Client Satisfaction Questionnaire CSQ-8, with 8 items, score 8-32. The higher the score, the more satisfied the patient is.

SECONDARY OUTCOMES:
Evolution of the patient's physical functions | Between the initial visit, the 3-month visit, and the 6-months visit
  Change in ALS-FRS-R (Amyotrophic lateral sclerosis functional rating scale revised) questionnaire score, score 0-48. The higher the score, the better the patient's physical function.
Non-inferiority of ventilatory efficiency compared to conventional management | Between the initial visit, the 3-month visit, and the 6-months visit
  Non-inferiority of efficiency will be assessed in a blinded manner by two third party experts in ventilation. This ventilatory efficiency will be assessed by S3-NIV (symptoms, sleep quality and side-effects related to the non-invasiv ventilation) questionnaire score 0-10. the higher the score, the fewer ALS-related symptoms the patient has.
Non-inferiority of ventilatory efficiency compared to conventional management | Between the initial visit, the 3-month visit, and the 6-months visit
  Non-inferiority of efficiency will be assessed in a blinded manner by two third party experts in ventilation. This ventilatory efficiency will be assessed by mean nocturnal oxygen saturation (SpO2, %) measured by oximetry
Non-inferiority of ventilatory efficiency compared to conventional management | Between the initial visit, the 3-month visit, and the 6-months visit
  Non-inferiority of efficiency will be assessed in a blinded manner by two third party experts in ventilation. This ventilatory efficiency will be assessed by time spent (in minutes) below 90% SpO2, measured by oximetry
Non-inferiority of ventilatory efficiency compared to conventional management | Between the initial visit, the 3-month visit, and the 6-months visit
  Non-inferiority of efficiency will be assessed in a blinded manner by two third party experts in ventilation. This ventilatory efficiency will be assessed by mean PtCO2 (in mmHg), measured by capnography
Non-inferiority of ventilatory efficiency compared to conventional management | Between the initial visit, the 3-month visit, and the 6-months visit
  Non-inferiority of efficiency will be assessed in a blinded manner by two third party experts in ventilation. This ventilatory efficiency will be assessed by time spent (in minutes) above 50 mmHg PtCO2 measured by capnography
Non-inferiority of ventilatory efficiency compared to conventional management | Between the initial visit, the 3-month visit, and the 6-months visit
  Non-inferiority of efficiency will be assessed in a blinded manner by two third party experts in ventilation. This ventilatory efficiency will be assessed by the treatment compliance (average daily use) through telemonitoring of the data recorded by the CPAP machine.
Non-inferiority of ventilatory efficiency compared to conventional management | Between the initial visit, the 3-month visit, and the 6-months visit
  Non-inferiority of efficiency will be assessed in a blinded manner by two third party experts in ventilation. This ventilatory efficiency will be assessed by the unintentional leakage through telemonitoring of the data recorded by the CPAP machine.
Non-inferiority of ventilatory efficiency compared to conventional management | Between the initial visit, the 3-month visit, and the 6-months visit
  Non-inferiority of efficiency will be assessed in a blinded manner by two third party experts in ventilation. This ventilatory efficiency will be assessed by the residual Apnea-Hypopnea Index (AHI) through telemonitoring of the data recorded by the CPAP machine.
The evolution of the efficiency of ventilation between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the initial visit, the 3-month visit, and the 6-months visit
  Comparison of the evolution of ventilation efficiency assessed from clinical parameters measured by S3-NIV (symptoms, sleep quality and side-effects related to the non-invasiv ventilation) questionnaire, score 0-10. the higher the score, the fewer ALS-related symptoms the patient has.
The evolution of the efficiency of ventilation between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the initial visit, the 3-month visit, and the 6-months visit
  Comparison of the evolution of ventilation efficiency assessed from mean PtCO2 (in mmHg), measured by capnography
The evolution of the efficiency of ventilation between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the initial visit, the 3-month visit, and the 6-months visit
  Comparison of the evolution of ventilation efficiency assessed from time spent (in minutes) below 90% SpO2, measured by oximetry
The evolution of the efficiency of ventilation between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the initial visit, the 3-month visit, and the 6-months visit
  Comparison of the evolution of ventilation efficiency assessed from mean nocturnal oxygen saturation (SpO2,%) measured by oximetry
The evolution of the efficiency of ventilation between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the initial visit, the 3-month visit, and the 6-months visit
  Comparison of the evolution of ventilation efficiency assessed from time spent (in minutes) above 50 mmHg PtCO2 measured by capnography
The evolution of the efficiency of ventilation between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the initial visit, the 3-month visit, and the 6-months visit
  Comparison of the evolution of ventilation efficiency assessed by the treatment compliance (average daily use) through telemonitoring of the data recorded by the CPAP machine.
The evolution of the efficiency of ventilation between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the initial visit, the 3-month visit, and the 6-months visit
  Comparison of the evolution of ventilation efficiency assessed by the unintentional leakage through telemonitoring of the data recorded by the CPAP machine.
The evolution of the efficiency of ventilation between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the initial visit, the 3-month visit, and the 6-months visit
  Comparison of the evolution of ventilation efficiency assessed by the residual Apnea-Hypopnea Index (AHI) through telemonitoring of the data recorded by the CPAP machine.
Patient satisfaction with teleconsultation itself (use and patient/doctor interaction) | After each teleconsultation (3-month visit and 6-month visit)
  Evaluation of the score of the Visit Satisfaction Questionnaire (VSQ-VF) score 0-100. The higher the score, the more satisfied the patient is.
The evolution of satisfaction between patients who have completed the teleconsultation follow-up visit and those who have completed the face-to-face follow-up visit | Between the 3-month visit, and the 6-months visit
  Comparison of the variation in the score of the visit satisfaction questionnaire, assessed by the VSQ-VF questionnaire, score 0-100. The higher the score, the more satisfied the patient is.
Physician satisfaction with teleconsultation | After each teleconsultation (3-month visit and 6-month visit)
  Evaluation made by Visual Analogue Scale (VAS) from 0 to 10 cm. The higher the score, the more satisfied the physician is.
Caregivers' satisfaction with the care of the relative | Between the initial visit, the 3-month visit, and the 6-months visit
  Change in caregiver satisfaction measured with client satisfaction questionnaire score (CSQ-8 modified) with 8 items, score 8-32. The higher the score, the more satisfied the caregivers' is.
The feasibility of home teleconsultation for ALS patients | Between the initial visit, the 3-month visit, and the 6-months visit
  Number of failed teleconsultations requiring rescheduling
Retention of follow-up modality | At 6 months
  Number of patients who changed follow-up modality, assessed by the number of face-to-face follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christel Saint-Raymond, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (2):
- France (2):
  - CHU Grenoble Alpes, Grenoble, France
  - CHU Montpellier, Montpellier, France